CLINICAL TRIAL: NCT06362499
Title: Effects of Unsupervised Inspiratory Muscle Training on Ventilation Variability in Post-covid-19 Patients: Protocol for Randomized Clinical Trial.
Brief Title: Effects of Unsupervised Inspiratory Muscle Training on Ventilation Variability in Post-covid-19 Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Patri-cia Angelica de Miranda Silva Nogueira, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2024-04-11; First posted 2024-04-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (GE) (Experimental): TMI with 30% of Pimax. with a weekly load increase of 10% of the Pimax value initial. The sessions will consist of 30 repetitions, 4 times a day, 2 sets in the morning and two sets in the afternoon, with a one-minute break between sets, 7 consecutive days a week, for 6 weeks. Individuals will be instructed to perform a rapid contraction of the inspiratory muscles and sustain it for 2 seconds, in each maneuver, and will have the possibility to rest after every 3 repetitions of the IMT, for 30 seconds, to avoid muscle fatigue or any other complications.
  Interventions: Device: Experimental Group
- Sham Group (SG) (Placebo Comparator): : Individuals will use a TMI device without any charge and will receive the same instructions as in G1. At the end of the research, the control group will be entitled to experimental treatment with the IMT protocol, if it proves to be effective.
  Interventions: Device: Experimental Group

INTERVENTIONS:
Device: Experimental Group — After the initial assessment, all volunteers will receive a POWERbreathe® classic light resistance device (POWERbreathe®, Nsc, Brazil), to carry out the training, and will be individually guided on how to use it and how to complete the protocol. They will perform a trial session to familiarize themselves with the device that will not be considered for analysis. Every week, volunteers will receive a telephone call from researcher 2, who will not participate in the evaluation, to confirm whether the exercise with the POWERbreathe® will be performed appropriately at the recommended frequency, intensity, and duration and whether there are any questions regarding the protocol. At the end of each week, participants will receive a video call from researcher 2 to adjust the device according to G1's weekly load progression.

SUMMARY:
Dysfunctional breathing and persistent hypocapnia can be associated with many of the symptoms experienced by patients such as dyspnea, fatigue, chest pain and palpitations. The identification of dysfunctional breathing and hypocapnia in these patients is important as it may represent a target for treatment.

In many of these patients, tachypnea at low levels of exertion suggests increased respiratory muscle activity, which can lead to the sensation of dyspnea. Sympathetic hyperactivity leads to excessive and irregular ventilation during exercise. In this way, inspiratory muscle training can improve symptoms (dysfunctional breathing), possibly by attenuating the metaboreflex (vagal modulation-attenuation of the sympathetic response) of the inspiratory muscle in post-covid-19 subjects, reducing ventilatory variability.

DETAILED DESCRIPTION:
Primary objective To evaluate the effects of an unsupervised inspiratory muscle training (IMT) protocol on the behavior of ventilatory variability.

Secondary objective Evaluate the effects of IMT on, respiratory muscle strength, pulmonary function, quality of life, peripheral muscle strength, functional capacity and adverse effects and adherence.

Material and methods Type of study and location of research This randomized, controlled, double-blind, parallel, two arm clinical trial will be conducted at the Laboratory of Health Assessment Measures (LABMAS), Department of Physiotherapy of the Federal University of Rio Grande do Norte (UFRN).

I The subjects included in the research will undergo three assessment stages: pre-training (Initial), post-training (6 weeks). Assessments in the pre-training period will be carried out in 1 day. After recruitment, participants will be invited to attend the UFRN Physiotherapy Department to carry out the first day of assessment by a previously trained evaluator blind to the intervention allocation group and will include anamnesis and physical examination, with measurement of vital signs. , anthropometric measurements, spirometry, respiratory muscle strength (manovacuometry), functional capacity (6-minute step test) and analysis of ventilatory variability (portable ventilator), assessment of peripheral muscle strength (dynamometry), quality of life (SF-36) .

The sample will be automatically randomized through the website www.randomization.com and allocated into two distinct groups: Experimental Group (GE): inspiratory muscle training and Sham Group (G2): IMT without load. Three evaluators will participate in the research: researcher 1 will be responsible only for the evaluations, researcher 2 for respiratory muscle training with weekly load adjustment and researcher 3 for randomization. The study will be double-blind, as researcher 1 and participants will not be aware of the allocation of subjects into groups, nor of the effects of the intervention.

After the initial assessment, all volunteers will receive a POWERbreathe® classic light resistance device (POWERbreathe®, Nsc, Brazil), to carry out the training, and will be individually guided on how to use it and how to complete the protocol. They will perform a trial session to familiarize themselves with the device that will not be considered for analysis. Every week, volunteers will receive a telephone call from researcher 2, who will not participate in the evaluation, to confirm whether the exercise with the POWERbreathe® will be performed appropriately at the recommended frequency, intensity, and duration and whether there are any questions regarding the protocol. At the end of each week, participants will receive a video call from researcher 2 to adjust the device according to G1's weekly load progression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes will be included, with a diagnosis of COVID-19 confirmed by RT-PCR, aged over 18 years, without any underlying respiratory or cardiac disease and reduced respiratory muscle strength (≤100 cmH2O). Reduced inspiratory muscle strength will be defined using MIP.

Exclusion Criteria:

* Patients with conditions impairing assessments, health complications that justify interrupting data collection (e.g., syncope, intense chest pain, or cough with blood-tinged sputum), hospitalized due to exacerbation of clinical conditions, or requested to leave the study will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Ventilation variability and ventilation efficiency | before and after 6 weeks
  For the ventilatory variables, the slope and intercept of the VE/VCO2 relationship will be obtained by simple linear regression of the type: VE = a * V´CO2 +/- b, with "a" corresponding to the slope of the relationship and "b" the interception value, including data from the peak loading exercise (RAMOS et al., 2013). We will also evaluate two new ventilation parameters, the constant rate of CO2 output (CO2CR) and the ventilation efficiency (ηVE). The two new variables were recently described (MULLER; SARAIVA et al., 2021). Briefly, the CO2CR will be obtained in a similar way to that described for the oxygen consumption efficiency curve, that is, taking the 10th base logarithm of VE on the x-axis against VCO2 on the y-axis. This relationship results in a characteristic quadratic function in most cases. The parameter "b" of the linear part of the equation type VCO2 = a * VE + b * V´E + c is called CO2CR.

SECONDARY OUTCOMES:
Respiratory muscle strength | before and after 6 weeks
  Patients will use a nasal clip and remain seated comfortably in a chair with back support, hip angle of 90˚, upper limbs resting on legs, and feet on floor. To measure MIP, patients will perform maximal expiration until residual volume, place the mouthpiece, and perform a maximal inspiratory effort against an occluded airway, and sustain for a minimum of one second.To measure MEP, the patient will inspire close to total lung capacity, place the mouthpiece, and perform a maximal expiratory effort against the occluded airway, maintaining for at least one second (NEDER et al.,1999). Patients will be constantly encouraged by the researcher during the test.For data analysis, at least three reproducible maneuvers will be performed with variability lower than 20%; the highest value will be registered. References values for the Brazilian population will be calculated according to age and gender (NEDER et al., 1999).
Pulmonary function | before and after 6 weeks
  Pulmonary volume and capacity will be evaluated using a calibrated spirometer (Koko Digidoser model, Spide, Longmont, USA) in an acclimatized room. Patients will be advised to avoid large meals one hour before the test, food and drinks with caffeine for at least six hours before the test, and alcoholic drinks on the day of the test (ATS, 2019).The test will consist in performing an inspiratory maneuver until total lung capacity, followed by maximal and forced expiration to residual volume using the spirometer. Tests will be performed with patients seated and hips and ankles flexed at 90º. A minimum of three tests will be conducted with variation less than 5%; the highest forced expiratory volume in the first second and forced vital capacity obtained will be compared with predicted values for the Brazilian population (PEREIRA, et al., 2007).
Quality of life - Medical Outcomes Study 36-Item Short Health Form Survey (SF-36) | before and after 6 weeks
  The Medical Outcomes Study 36-Item Short Health Form Survey (SF-36) is a multidimensional questionnaire translated and validated for the Brazilian reality (CICONELLI et al., 1999; LAGUARDIA et al., 2011) that was developed to assess quality of life related to health. The instrument consists of 36 items, distributed in 8 domains that encompass two major components: the physical (physical aspects, bodily pain, general health status and physical function) and the mental (emotional aspects, social function, mental aspects and vitality). Scores range from 0 to 100 for each subscale, with higher scores indicating a better health-related quality of life (WARE; SHERBOURNE, 1992).
Peripheral muscle strength | before and after 6 weeks
  Handgrip strength will be measured using a hydraulic handheld dynamometer (Saehan1). Maximal isometric strength of the dominant hand will be assessed with patients seated comfortably in a chair, with knee and ankle joints at 90º, shoulder of dominant arm forward and in neutral rotation, elbow flexed at 90º near upper body, forearm in neutral position, and wrist between 0º to 30º of extension and 0º to 15º of ulnar deviation. Participants will be requested to perform maximal isometric strength for five seconds without moving other body parts (NOVAES et al., 2009). Three measurements will be performed with one-minute interval in between, and the average will be considered for analysis. Patients will be considered fragile if the average of three measurements is between 20% of lower distribution values, according to the World Health Organization (HOLAND et al., 2014).
Functional capacity | before and after 6 weeks
  Participants will perform the six-minute step test. They will be instructed to climb down the 20 cm step at a speed that allows them to perform the maximum number of steps in 6 minutes. They can start the test with any lower limb. The number of steps the participant takes will be counted at the end of the test (a cycle of going up and down will be considered as one step). Before and after the test, heart rate (HR) will be assessed (Polar Vantage NVTM, model 1901001, Oulu, Finland), blood pressure and SpO2, dyspnea and lower limb fatigue will be questioned using a modified Borg scale (0-10). Two tests will be carried out with an interval of 30 minutes between them and the values of the variables obtained in the best test, that is, the test in which the individual climbs the greatest number of steps will be used for analysis (ALBUQUERQUE et al., 2022).
Adverse effects and adherence | before and after 6 weeks
  Adverse effects and adherence will be assessed using a training diary will be given to all patients to assess adverse effects and adherence. After all training sessions, they will be encouraged to fill the diary, registering positive and negative observations and complications during and after training. Adherence will be assessed considering every time patients register the realization of the session. Fulfilled sessions will be added and then divided by the total number of sessions patients could perform.
  Adherence to training will be considered by verifying the number of days that patient performed the sessions. The sum of all sessions performed will be divided by the total number of sessions that patients must perform. Adverse effects will consider all complications registered in the diary or mentioned during final evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Nogueira, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (2):
- Brazil (2):
  - Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte
  - Patrícia Nogueira, Natal, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No